CLINICAL TRIAL: NCT01337089
Title: A Multicenter, Non-comparative, Open-label Extension Study to Assess the Long Term Safety of Sativex® Oromucosal Spray (Sativex®; Nabiximols) as Adjunctive Therapy in Patients With Uncontrolled Persistent Chronic Cancer Related Pain
Brief Title: Long Term Safety of Sativex Oromucosal Spray (Sativex®; Nabiximols) as Adjunctive Therapy in Patients With Uncontrolled Persistent Chronic Cancer Related Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWCA0999; 2009-016529-32 (EudraCT Number)
Record Dates: First submitted 2011-04-12; First posted 2011-04-18 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Pain; Advanced Cancer
Keywords: Cancer pain; Opioid therapy; Inadequate analgesia; Optimized chronic opioid therapy
MeSH Terms: conditions — Pain; Cancer Pain | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non-comparative, open-label Nabiximols (Experimental): Nabiximols was self-administered by participants as a 100 microliter (μL) oromucosal spray, in the morning and evening, up to a maximum of 10 sprays per day for 6 months. Nabiximols oromucosal spray contained delta-9-tetrahydrocannabinol (THC) (27 milligrams [mg]/milliliter [mL]):cannabidiol (CBD) (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD.
  Interventions: Drug: Nabiximols

INTERVENTIONS:
Drug: Nabiximols
  Other Names: Sativex®

SUMMARY:
This was a six-month open-label extension (OLE) study to evaluate the safety of long-term nabiximols (Sativex®) therapy when used as an adjunctive treatment in participants with advanced cancer. The study provided continued availability of nabiximols to participants who completed a preceding Phase 3 study and new (de novo) participants.

DETAILED DESCRIPTION:
This was a 6-month, multicenter, non-comparative, OLE study to evaluate the safety of long-term nabiximols use as an adjunctive measure in participants with advanced cancer. The study provided continued availability of nabiximols to participants who completed a preceding double-blind phase 3 study and de novo participants. Consenting eligible participants entered the extension study (Day 1) on the same day as the "end of treatment" visit of a parent study or within 7 days of the "end of treatment" visit or on the day of the "safety follow-up visit" of the parent study. The "safety follow-up" visit of a parent study was performed on the same day as Day 1, if the participant did not enter the OLE study on the same day as the "end of treatment" visit of a parent study. De novo participants attended a screening visit 3 to 14 days prior to enrollment (Day 1). All participants commenced dosing on Day 1. Further study visits took place after 2 weeks (Day 15), and every 4 weeks thereafter until the end of treatment period on Day 183 or earlier if the participant withdrew from the study.

Treatment was started as a single spray in the evening on the first day (Day 1). Participants then gradually titrated by 1 additional spray per day to an individualized dose, balancing efficacy and tolerability. Participants had to complete titration within 14 days of their first dose of study drug and then continue at the same dose for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant had completed the parent study within the last seven days
* Willing and able to give written informed consent
* Willing and able to comply with all study requirements

Exclusion Criteria:

* The participant was using cannabis or cannabinoid based medications, other than the parent study investigational medicinal product (IMP), and was unwilling to abstain for the duration of the study
* Any history or immediate family history of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition
* Any known or suspected history of a substance abuse/dependence disorder (including opiate abuse/dependence prior to the diagnosis of cancer), current heavy alcohol consumption (more than 60 grams [g] of pure alcohol per day for men, and more than 40 g of pure alcohol per day for women), current use of an illicit drug or current non-prescribed use of any prescription drug
* Had poorly controlled epilepsy or recurrent seizures (for example, one or more seizure during the last year)
* Had experienced myocardial infarction or clinically significant cardiac dysfunction within the last 12 months or had a cardiac disorder that, in the opinion of the investigator would have put the participant at risk of a clinically significant arrhythmia or myocardial infarction
* Had significantly impaired renal function
* Had significantly impaired hepatic function at the "end of treatment" visit of the parent study
* Female participants of child-bearing potential and male participants whose partner was of child-bearing potential, unless willing to ensure that they or their partner used effective contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for 3 months thereafter (however, a male condom should not have been used in conjunction with a female condom as this may not have proven effective)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2011-01-19 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2016-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (119):
- United States (34):
  - Phoenix, Arizona
  - El Cajon, California
  - Gilroy, California
  - Glendale, California
  - Santa Rosa, California
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Holiday, Florida
  - Jacksonville, Florida
  - Lynn Haven, Florida
  - Miami, Florida
  - Stuart, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Marietta, Georgia
  - Newnan, Georgia
  - Stockbridge, Georgia
  - Woodlawn, Illinois
  - Ashland, Kentucky
  - Bossier City, Louisiana
  - Shreveport, Louisiana
  - Saint Louis Park, Minnesota
  - Kansas City, Missouri
  - Missoula, Montana
  - Berlin, New Jersey
  - New York, New York
  - Flat Rock, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Laredo, Texas
  - Salt Lake City, Utah
  - Lacey, Washington
- Parkville, Australia
- Brussels, Belgium
- Bulgaria (3):
  - Gabrovo
  - Varna
  - Vratsa
- Czechia (9):
  - Benešov
  - České Budějovice
  - Jablonec nad Nisou
  - Most
  - Nová Ves pod Pleší
  - Ostrava
  - Pilsen
  - Sokolov
  - Teplice
- Germany (7):
  - Berlin
  - Frankfurt
  - Jena
  - Lünen
  - Stadtroda
  - Wetzlar
  - Wiesbaden
- Hungary (6):
  - Deszk
  - Komárom
  - Miskolc
  - Nyíregyháza
  - Szekszárd
  - Szikszó
- Israel (4):
  - Beersheba
  - Haifa
  - Ramat Gan
  - Ẕerifin
- Italy (3):
  - Garbagnate Milanese
  - Piacenza
  - Torino
- Latvia (2):
  - Rēzekne
  - Riga
- Lithuania (3):
  - Klaipėda
  - Šiauliai
  - Vilnius
- Mexico (2):
  - Chihuahua City
  - Distrito Federal
- Poland (14):
  - Bialystok
  - Bielsko-Biala
  - Bydgoszcz
  - Czeladź
  - Częstochowa
  - Działdowo
  - Gdansk
  - Gliwice
  - Kłodzko
  - Opole
  - Ostrowiec Świętokrzyski
  - Poznan
  - Warsaw
  - Włocławek
- Puerto Rico (2):
  - Ponce
  - San Juan
- Romania (13):
  - Baia Mare
  - Brăila
  - Bucharest
  - Cluj-Napoca
  - Constanța
  - Craiova
  - Focşani
  - Iași
  - Oradea
  - Satu Mare
  - Sibiu
  - Suceava
  - Târgovişte
- Granada, Spain
- Taiwan (2):
  - Taichung
  - Tainan
- United Kingdom (12):
  - Bury
  - Bury St Edmunds
  - Cheltenham
  - Crumpsall
  - Edinburgh
  - Gorleston-on-Sea
  - Leeds
  - Manchester
  - Norwich
  - Plymouth
  - Weston-super-Mare
  - Withington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled in this study included those who had taken part in studies NCT01262651 (GWCA0958), NCT01361607 (GWCA0962), and NCT01424566 (GWCA1103) and who chose to continue treatment by enrolling in this study, as well as new (de novo) participants who met all inclusion criteria and did not meet any of the exclusion criteria.
Pre-assignment Details: For the de novo participants enrolled in this study, a screening visit took place 3 to 14 days prior to enrollment.
Groups:
- Nabiximols: Nabiximols was self-administered by participants as a 100 microliter (μL) oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day, for 6 months. Nabiximols oromucosal spray contained delta-9-tetrahydrocannabinol (THC) (27 milligram [mg]/milliliter [mL]):cannabidiol (CBD) (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD.
Period: Overall Study
Arm/Group | Nabiximols
Started | 660
Received at Least 1 Dose of Study Drug | 660
Safety Population | 660
Efficacy Dataset | 659 (One participant withdrew after administering nabiximols, but no efficacy data were collected.)
Completed | 256
Not Completed | 404
Not completed — Adverse Event | 237
Not completed — Withdrawal by Subject | 129
Not completed — Withdrawal by Investigator | 33
Not completed — Met Withdrawal Criteria | 3
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least 1 dose of nabiximols.
Groups:
- Nabiximols: Nabiximols was self-administered by participants as a 100 μL oromucosal spray in the morning and evening, up to a maximum of 10 sprays per day, for 6 months. Nabiximols oromucosal spray contained THC (27 mg/mL):CBD (25 mg/mL), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavoring. Each 100 μL actuation delivered 2.7 mg THC and 2.5 mg CBD.
Arm/Group | Nabiximols
Number analyzed (Participants) | 660
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 313
  Male | 347

OUTCOME MEASURES:

1. Primary Outcome: Percent Of Participants With Treatment-emergent Adverse Events
Description: Treatment-emergent Adverse Events (TEAEs) were coded according to the Medical Dictionary for Regulatory Activities (MedDRA) dictionary version 17.0. A TEAE is defined as an adverse event with an onset after the start of study drug treatment. The percent of participants who experienced one or more TEAEs is reported.
Time Frame: Baseline, Day 183
Population: The Safety Population included all participants receiving at least 1 dose of study drug.
Measure: Number; unit: percent of participants
Arm/Group | Nabiximols
Number analyzed (Participants) | 660
percent of participants | 82.9

2. Secondary Outcome: Change From Baseline In Mean NRS Average Pain During The Last Period
Description: Participants indicated the level of pain experienced in the last 24 hours on an 11-point Numerical Rating Scale (NRS), where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine." Change in mean NRS average pain was calculated as: Last Period NRS average pain score - Baseline NRS average pain score.
  A negative value indicates an improvement in average pain score from Baseline.
Time Frame: Baseline, Last Period (Days 156-183) or last 27 days of treatment
Population: The Safety Population included all participants receiving at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nabiximols
Number analyzed (Participants) | 634
units on a scale | 0.0 (1.8)

3. Secondary Outcome: Change From Baseline In Mean Sleep Disruption NRS During The Last Period
Description: Participants indicated the level of sleep disruption experienced in the last 24 hours on an 11-point NRS, where a score of 0 indicated "did not disrupt sleep" and a score of 10 indicated "completely disrupted (unable to sleep at all)." Change in mean sleep disruption NRS was calculated as: Last Period sleep disruption NRS score - Baseline sleep disruption NRS score.
  A negative value indicates an improvement in sleep disruption score from Baseline.
Time Frame: Baseline, Last Period (Days 156-183) or last 27 days of treatment
Population: The Safety Population included all participants receiving at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nabiximols
Number analyzed (Participants) | 634
units on a scale | 0.1 (1.9)

4. Secondary Outcome: Patient Satisfaction Questionnaire At Last Visit (Up To Day 183)
Description: The Patient Satisfaction Questionnaire (PSQ) was used to assess level of satisfaction of the participant with the study drug, with the markers "extremely satisfied, very satisfied, slightly satisfied, neutral, slightly dissatisfied, very dissatisfied, extremely dissatisfied". Last visit refers to the last visit that a participant completed the assessment.
Time Frame: Last Visit (up to Day 183)
Population: The Safety Population included all participants receiving at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Nabiximols
Number analyzed (Participants) | 618
Participants
  Extremely Satisfied | 56
  Very Satisfied | 230
  Slightly Satisfied | 185
  Neutral | 82
  Slightly Dissatisfied | 33
  Very Dissatisfied | 22
  Extremely Dissatisfied | 10

5. Secondary Outcome: Change From Baseline In NRS Constipation At Last Visit (Up To Day 183)
Description: Participants indicated level of constipation on an 11-point NRS, where a score of 0 was "no constipation", and 10 was "constipation as bad as you can imagine." Last visit refers to the last visit that a participant completed the assessment.
  Change in NRS constipation score was calculated as: Last Visit NRS constipation score - Baseline NRS constipation score.
  A negative value indicates improvement in condition from Baseline.
Time Frame: Baseline, Last Visit (up to Day 183)
Population: The Safety Population included all participants receiving at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nabiximols
Number analyzed (Participants) | 619
units on a scale | -0.1 (2.5)

ADVERSE EVENTS:
Time Frame: Up to Day 197 post-enrollment
Arm/Group | Nabiximols
Serious Adverse Events (participants affected / at risk) | 301/660
Other Adverse Events (participants affected / at risk) | 291/660
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nabiximols (N=660)
Anaemia (Blood and lymphatic system disorders) | 8
Anaemia Of Malignant Disease (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Angina Pectoris (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Cardiopulmonary Failure (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 3
Pyloric Stenosis (Congenital, familial and genetic disorders) | 1
Deafness Neurosensory (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenal Insufficiency (Endocrine disorders) | 1
Blindness (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 7
Abdominal Pain (Gastrointestinal disorders) | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis Erosive (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Intestinal Obstruction (Gastrointestinal disorders) | 1
Mechanical Ileus (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2
Tongue Haemorrhage (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 4
Device Occlusion (General disorders) | 1
General Physical Health Deterioration (General disorders) | 1
Local Swelling (General disorders) | 1
Pain (General disorders) | 6
Pyrexia (General disorders) | 3
Gastroenteritis (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Catheter Site Infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Clostridium Difficile Colitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Klebsiella Sepsis (Infections and infestations) | 1
Lobar Pneumonia (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 4
Pelvic Abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pseudomembranous Colitis (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1
Staphylococcal Sepsis (Infections and infestations) | 1
Subacute Endocarditis (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 5
Femur Fracture (Injury, poisoning and procedural complications) | 1
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1
Procedural Headache (Injury, poisoning and procedural complications) | 2
Radiation Oesophagitis (Injury, poisoning and procedural complications) | 1
Shunt Occlusion (Injury, poisoning and procedural complications) | 1
Stoma Complication (Injury, poisoning and procedural complications) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 4
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 209
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases To Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/313
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spinal Cord Compression (Nervous system disorders) | 3
Altered State Of Consciousness (Nervous system disorders) | 1
Balance Disorder (Nervous system disorders) | 1
Carotid Artery Stenosis (Nervous system disorders) | 1
Cerebral Infarction (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 3
Grand Mal Convulsion (Nervous system disorders) | 1
Dementia With Lewy Bodies (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Completed Suicide (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 4
Mental Status Changes (Psychiatric disorders) | 2
Suicide Attempt (Psychiatric disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 5
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Genital Haemorrhage (Reproductive system and breast disorders) | 1
Vaginal Fistula (Reproductive system and breast disorders) | 1/313
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 1
Dry Gangrene (Skin and subcutaneous tissue disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 4
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Inferior Vena Caval Occlusion (Vascular disorders) | 1
Venous Thrombosis Limb (Vascular disorders) | 1
Convulsion (Nervous system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nabiximols (N=660)
Anaemia (Blood and lymphatic system disorders) | 39
Nausea (Gastrointestinal disorders) | 86
Vomiting (Gastrointestinal disorders) | 59
Constipation (Gastrointestinal disorders) | 44
Diarrhoea (Gastrointestinal disorders) | 41
Fatigue (General disorders) | 35
Decreased Appetite (Metabolism and nutrition disorders) | 49
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 41
Dizziness (Nervous system disorders) | 51
Somnolence (Nervous system disorders) | 38
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37
Asthenia (General disorders) | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days